CLINICAL TRIAL: NCT05081921
Title: A Randomized, Double Blind, Two Arms, Controlled Phase I/II Safety and Efficacy Study on MesoCellA-Ortho Tissue Engineered Product Intraarticularly Administrated in Adult Patients With Osteoarthrosis
Brief Title: Clinical Trial to Evaluate Safety and Efficacy of MesoCellA-Ortho Tissue-Engineered Advanced Therapy Product in Patients With Osteoarthrosis and Civilisation Diseases
Acronym: BioMiStem-CT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Collaborators: National Center for Research and Development, Poland (Other); KCRI (Other)
Responsible Party: Principal Investigator, Prof. Krzysztof FICEK, MD, PhD, DSc, Professor, Galen Ortopedia Sp. z o. o
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JU-BioMiStem-01; 2019-005000-17 (EudraCT Number)
Record Dates: First submitted 2021-08-23; First posted 2021-10-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis of Knee
Keywords: Osteoarthritis; Mesenchymal stem cells; Autologous stem cells; Adipose tissue; Type 2 diabetes; Obesity; Civilisation diseases
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomization list and envelope based procedure will be used to eliminate selection bias. In order to maximally reduce bias, the trial is double-blind, with all involved subjects and the investigator blinded to the treatment. The randomization list will not be available to any person involved in the conduct. The evaluation of the trial results will not be performed until the trial database is locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- MesoCellA-Ortho - treated Patients with type 2 diabetes and with obesity (Experimental): The patients with osteoarthritis of knee, suffering also with type 2 diabetes and obesity (BMI > 30) will be enrolled into this group and will be treated with MesoCellA-Ortho (single intraarticular application of 20 mln of AT-MSCs resuspended in carrier solution mixed with hyaluronic acid)
  Interventions: Drug: MesoCellA-Ortho administration
- Control Patients with type 2 diabetes and obesity (Active Comparator): The patients with osteoarthritis of knee, suffering also with type 2 diabetes and obesity (BMI > 30) will be enrolled into this group and will be injected with hyaluronic acid (single intraarticular application of HA)
  Interventions: Drug: HA administration
- MesoCellA-Ortho - treated Patients without type 2 diabetes and with obesity (Experimental): The patients with osteoarthritis of knee, suffering also with obesity (BMI > 30), but with no type 2 diabetes will be enrolled into this group and will be treated with MesoCellA-Ortho (single intraarticular application of 20 mln of AT-MSCs resuspended in carrier solution mixed with hyaluronic acid)
  Interventions: Drug: MesoCellA-Ortho administration
- Control Patients without type 2 diabetes and with obesity (Active Comparator): The patients with osteoarthritis of knee, suffering also with obesity (BMI > 30), but with no type 2 diabetes will be enrolled into this group and will be injected with hyaluronic acid (single intraarticular application of HA)
  Interventions: Drug: HA administration
- MesoCellA-Ortho - treated Patients without type 2 diabetes and without obesity (Experimental): The patients with osteoarthritis of knee, with no obesity (BMI < 30) nor type 2 diabetes will be enrolled into this group and will be treated with MesoCellA-Ortho (single intraarticular application of 20 mln of AT-MSCs resuspended in carrier solution mixed with hyaluronic acid)
  Interventions: Drug: MesoCellA-Ortho administration
- Control Patients without type 2 diabetes and without obesity (Active Comparator): The patients with osteoarthritis of knee, with no obesity (BMI < 30) nor type 2 diabetes will be enrolled into this group and will be injected with hyaluronic acid (single intraarticular application of HA)
  Interventions: Drug: HA administration

INTERVENTIONS:
Drug: MesoCellA-Ortho administration — Single dose of MesoCellA-Ortho product consisting of 20 mln of autologous adipose tissue-derived mesenchymal stem/ stromal cells (AT-MSCs) will be administrated intraarticularly in patients enrolled in "MesoCellA-Ortho- treated" groups.
  Other Names: Experimental treatment
  Arms: MesoCellA-Ortho - treated Patients with type 2 diabetes and with obesity; MesoCellA-Ortho - treated Patients without type 2 diabetes and with obesity; MesoCellA-Ortho - treated Patients without type 2 diabetes and without obesity
Drug: HA administration — Single dose of hyaluronic acid (HA) will be administrated intraarticularly as an active control in patients enrolled in "Control Patients" groups.
  Other Names: Standard treatment (control)
  Arms: Control Patients with type 2 diabetes and obesity; Control Patients without type 2 diabetes and with obesity; Control Patients without type 2 diabetes and without obesity

SUMMARY:
The aim of the study is to evaluate safety, tolerability and clinical efficacy of a newly developed MesoCellA-Ortho tissue-engineered advanced therapy medicinal product in adult patients suffering with osteoarthritis and additionally burdened with other civilisation diseases such as type 2 diabetes and/ or obesity.

The active substance of MesoCellA-Ortho consists of in vitro expanded autologous human adipose tissue-derived mesenchymal stem/ stromal cells (AT-MSCs) resuspended in carrier solution for intraarticular injections for individual patents.

DETAILED DESCRIPTION:
To evaluate safety, tolerability and clinical efficacy of a MesoCellA-Ortho product, the active substance of MesoCellA-Ortho consisting of 20 mln in vitro expanded autologous human adipose tissue-derived mesenchymal stem/ stromal cells (AT-MSCs) will be intraarticularly administrated in adult patients with osteoarthritis and additionally burdened with other civilisation diseases such as type 2 diabetes and/ or obesity. Hyaluronic acid (HA) will be used as a Control.

The safety and clinical outcome of the treatment will be evaluated during 6 months of followup, considering patient's subjective pain level and evaluation of the improvement of knee joint function.

ELIGIBILITY:
Inclusion Criteria:

1. Knee cartilage lesions (osteoarthritis II/III grade in Kellgren-Lawrence scale confirmed in X-ray)
2. Age between 40-70 years (inclusive)
3. No contraindications for liposuction
4. No contraindications for the general use of biological treatment, stem cells, PRP and whole autologous blood
5. Availability to take part into all study visits, barring unforeseen circumstances
6. Able and willing to perform exercises at home given by a physiotherapist
7. Contraceptive (birth control pills, injection, pessary or intrauterine device (IUD), spermicide condoms)
8. The pain intensity in treated knee not lower than grade 3 (on 11-point Numerical Rating Scale)

Exclusion Criteria:

1. A history of cancer for 2 years before screening. In case of history of cancer medical above 2 years, consultation with oncologist and her/his permission for participation in clinical trial will be obligatory.
2. Pregnant or breastfeeding women.
3. Allergy or poor tolerance of hyaluronic acid.
4. Diabetes mellitus type 1, diabetes mellitus type 2 on insulin treatment.
5. Lack of medical consultation in case of patients with diabetes group.
6. Comorbidities significantly affecting overall health (e.g. history of myocardial infarction, heart failure, thrombophlebitis, arterial hypertension (hypertensive crises), chronic obstructive pulmonary disease, renal failure, liver failure, advanced atherosclerosis, psychoorganic syndrome, hemiparesis, history of stroke).
7. Current or medical history of the patient: inflammatory diseases of the joints (e.g. gout, reactive arthritis, psoriatic arthritis, seronegative arthritis involving the spine joints, septic arthritis, prior diagnosis of target arthrosis with crystal precipitation or elevated CRP in the condition, inflammation), osteonecrosis, osteoporotic fractures or other painful joint diseases other than osteoarthritis; secondary causes of osteoarthritis (e.g. rheumatoid arthritis, fibromyalgia, birth defects).
8. Current or medical history of the patient concerning carrier state or diseases: HIV, syphilis, HBV, HCV, EBV.
9. Symptomatic sciatica with radiation of pain to the examined limb.
10. Symptomatic osteoarthritis of the hip of both limbs.
11. Significant knee injuries within 6 months such as: ligament injuries, distal femur fracture or proximal tibia fracture, arthrofibrosis or cyclops lesions.
12. Endoprosthesis of the hip or knee joints.
13. Partial / total knee or hip joints replacement planned during the study.
14. Surgical operation of the lower limbs (including arthroscopy) within 6 months before screening visit or planned during the study.
15. Constant use of orthopaedic aids.
16. Intolerance or hypersensitivity to any component of the preparation.
17. Use of alternative treatment methods i.e. acupuncture within 4 weeks before screening visit or planning their use during the study.
18. Use in the treatment of osteoarthritis:

    * Hyaluronates (injections - test knee) within 3 months
    * Corticosteroids (injections) within 3 months
    * Oral corticosteroids within 3 months
19. If available, recent (<14 days) blood tests results outside of the allowable ranges (e. g. morphology, electrolytes, blood clotting APTT, INR, fibrinogen, CRP, glucose) if significant for participation in clinical study, particularly regarding contraindication for liposuction procedure.
20. If available, positive results of laboratory blood tests (HIV, syphilis, HBV, HCV, CMV -IgM antibodies, mycoplasmas -IgM antibodies, toxoplasmosis IgM antibodies, EBV IgM antibodies) if significant for participation in clinical study, particularly regarding contraindication for liposuction procedure.
21. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.
22. Known allergic reactions to antibiotics used in cell culture: penicillin, streptomycin, amphotericin B.
23. Intolerance or hypersensitivity to any of the anesthetics (including lignocaine).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Nature, incidence and severity of adverse events (AEs) | Month 6 Follow-up
  The measure of safety used in this study are routine clinical procedures. They include a close vigilance for, and stringent reporting of selected local and systemic reactions, adverse events including serious adverse events.
  After 4th rehabilitation visit to study termination, only AEs of special interest and serious adverse events (SAEs), AEs leading to withdrawal from the study and concomitant medications used to treat adverse events will be collected. The AEs of special interest related directly to the state of the knee after intraarticular administration will be: excessive warming of the knee, pain, suffusion, hematoma, knee locking, decrease ROM.
  The prevalence, duration and severity of AEs of special interest will be additionally analyzed in the study.
Change in Numerical Rating Scale (NRS) | Month 3 and Month 6 Follow-up
  The numerical scale is one of the most commonly used pain scales in medicine. The NRS consists of a numeric version of the visual analog scale. It is labeled from 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable". This scale can help guide the diagnostic process, track the progression of the pain, and more.
  Patients will report intensity of pain only in knee subjected to the treatment in the study.
Change in joint swelling | Month 3 and Month 6 Follow-up
  Evaluation the joint swelling during physical examination by 4-items scale: none, mild, moderate, severe. Joint swelling will be assessed only knee subjected to the treatment in the study.
Change in the 36-Item Short Form Survey (SF-36) | Month 6 Follow-up
  SF-36 is an oft-used, well-researched, self-reported measure of health. The SF-36 is often used as a measure of a person or population's quality of life. It comprises 36 questions which cover eight domains of health: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); 8) general health perceptions.
Change in Knee injury and Osteoarthritis Outcome Score (KOOS) | Month 3 and Month 6 Follow-up
  Change in Knee injury and Osteoarthritis Outcome Score (KOOS). It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL)
  The five patient-relevant subscales of KOOS are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic assessment scales and generic measures.
  Only knee subjected to treatment will be evaluated by KOOS survey.
Change in the International Knee Documentation Committee (IKDC 2000) | Month 3 and Month 6 Follow-up
  Change in IKDC Questionnaire score. The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee. Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function The transformed score is interpreted as a measure of function such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with activities of daily living or sports activities and the absence of symptoms.
  Only knee subjected to treatment will be evaluated by IKDC 2000 survey.

SECONDARY OUTCOMES:
Change in cartilage morphology | Month 6 Follow-up
  Cartilage morphology on MRI. Change in the modified Outerbridge (Modified Outerbridge classification of cartilage defects) classification. It is based on grading cartilage lesions, in which lesions are graded: 0 - normal cartilage, 1 - signal intensity alterations with an intact surface of the articular cartilage compared with the surrounding normal cartilage, 2 - partial thickness defect of the cartilage, 3 - fissuring of the cartilage to the level of the subchondral bone, 4 - exposed subchondral bone.
  Only knee subjected to treatment will be evaluated by MRI.
Change in cartilage T2 relaxation time mapping in MRI | Month 6 Follow-up
  Measurement of relaxation time (measured in milliseconds, ms) in selected ROIs (Region of Interest) in both medial and lateral femoral and tibial condyle. There will be: 6 ROIs in medial femoral condyle, 6 ROIs in lateral femoral condyle, 4 ROIs in medial tibia, and 4 ROIs in lateral tibia.
  Only knee subjected to treatment will be evaluated by MRI.
Changes in bone marrow edema-like lesions (BMLs) | Month 6 Follow-up
  The occurrence of bone marrow edema-like lesions (BMLs) in MRI will be checked. If bone marrow edema-like lesion is present then measurements of width and length (mm) in: medial femoral condyle, lateral femoral condyle, medial tibia, lateral tibia will be performed.
  Only knee subjected to treatment will be evaluated by MRI. It is hypothesized that the size of BMLs should decrease in second MRI.
Change in weight distribution on stable platform | Month 6 Follow-up
  Weight distribution on stable platform will be performed for objective evaluation of lower limb loading symmetry during 5 exercises: standing, standing with eyes closed, calf raises, squat, jump. Minimum, maximum and average weight-bearing value (measured in kilograms, kg) of the left and right lower extremity will be recorded.
  It is expected that predicted lower limb loading asymmetry in patients will transform to symmetry after MSCs treatment and rehabilitation.
Change in Range of motion (ROM) | Month 6 Follow-up
  Measurement of knee flexion and extension angles (in degrees, °). Normal ROM at the knee is considered to be 0 degrees of extension (completely straight knee joint) to 135 degrees of flexion (fully bent knee joint).
  Knee flexion angle, knee extension angle, knee hyperextension (if yes, hyperextension angle), hip range of motion (normal/abnormal) will be evaluated in left and right lower extremity.
Change in ultrasonographic findings in knee joint | Month 3 and Month 6 Follow-up
  During ultrasound examination, the volume of effusion (mL) will be assessed. The lateral and medial meniscus, lateral and medial knee, and patellofemoral joint will be evaluated (normal/abnormal; if abnormal, details are needed).

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Ficek, Prof., MD, PhD, DSc, Principal Investigator — Galen Ortopedia Sp. z o. o
Locations (1):
- Galen - Ortopedia Sp. Z O.O., Bieruń, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided